CLINICAL TRIAL: NCT00778050
Title: A Relative Bioavailability Study of 600 mg Amoxicillin Dispersible Tablets vs 400 mg/ 5 mL Amoxil ® for Oral Suspension Under Fasting Conditions.
Brief Title: Bioequivalence Study of Amoxicillin Dispersible 600 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R02 - 914
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence, amoxicillin 600mg fasting conditions
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): amoxicillin tablets for oral suspension 600 mg by Ranbaxy Laboratories Limited
  Interventions: Drug: Amoxicillin 600mg
- 2 (Active Comparator): Amoxil ® for oral suspension 400 mg/ 5 mL by SmithKline Beecham Pharmaceuticals (600mg dose)
  Interventions: Drug: Amoxicillin 600mg

INTERVENTIONS:
Drug: Amoxicillin 600mg

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of amoxicillin tablets for oral suspension 600 mg by Ranbaxy Laboratories Limited with that of Amoxil ® for oral suspension 400 mg/ 5 mL by SmithKline Beecham Pharmaceuticals following single oral dose (600 mg) in healthy, adult, subjects under fasting conditions using a randomized two-way crossover design.

DETAILED DESCRIPTION:
A single oral dose of the test or reference product was administered to volunteers on two separate occasions under fasting conditions with at least a 7 day washout between the doses. Twenty-six healthy volunteers were randomly assigned to the test or the reference products. Food and fluid intake were controlled during each confinement period.

Twenty six (26) healthy subjects (16 males and 10 females) were enrolled in the study, of which 25 subjects completed the clinical phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. All volunteers selected for this study will be healthy men or women 18 years of age or older at the time of dosing
2. The weight range will not exceed ± 20% for height and body frame as per Desirable Weights for Adults - 1983 Metropolitan Height and Weight Table
3. Each volunteer will complete a screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures
4. If female and:

   * of child bearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or
   * is postmenopausal for at least 1 year; or
   * is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

1. Volunteers with a recent history of drug or alcohol addiction or abuse
2. Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigators)
3. Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
4. Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen
5. Volunteers demonstrating a positive drug abuse screen when screened for this study
6. Female volunteers demonstrating a positive pregnancy screen
7. Female volunteers who are currently breastfeeding
8. Volunteers with a history of allergic response(s) to amoxicillin or related drugs
9. Volunteers with a history of clinically significant allergies including drug allergies
10. Volunteers with a clinically significant illness during the 4 weeks prior to period I dosing (as determined by the clinical investigators)
11. Volunteers who currently use tobacco products
12. Volunteers who have taken any drug known o induce or inhibit hepatic drug metabolism in the 30 days prior to period I dosing
13. Volunteers who report donating greater than 150 mL of blood within 30 days prior to period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
14. Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
15. Volunteers who report receiving any investigational drug within 30 days prior to period I dosing
16. Volunteers who report taking any systemic prescription medication in the 14 days prior to period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-10; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute Ltd., Fargo, North Dakota, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html